CLINICAL TRIAL: NCT00072540
Title: S0212: Phase IIb Randomized Study of Celecoxib in Patients With High-Grade Squamous Intraepithelial Lesions of the Cervix
Brief Title: S0212 Celecoxib in Treating Patients With High-Grade Squamous Intraepithelial Lesions of the Cervix
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: drug issues
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000340176; S0212 (Other: SWOG); U10CA037429 (NIH)
Record Dates: First submitted 2003-11-04; First posted 2003-11-05 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Stage 0 Cervical Cancer; High-grade Squamous Intraepithelial Lesion
MeSH Terms: conditions — Uterine Cervical Dysplasia; Squamous Intraepithelial Lesions | interventions — Celecoxib; Biological Therapy; Chemoprevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: celecoxib
Procedure: anti-cytokine therapy
Procedure: antiangiogenesis therapy
Procedure: biological therapy
Procedure: cancer prevention intervention
Procedure: chemoprevention of cancer
Procedure: enzyme inhibitor therapy
Procedure: growth factor antagonist therapy

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development of cancer. Celecoxib may be effective in preventing cervical cancer.

PURPOSE: Randomized phase II trial to study the effectiveness of celecoxib in preventing cervical cancer in patients who have high-grade squamous intraepithelial lesions of the cervix.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the complete response rate in patients with high-grade squamous intraepithelial lesions of the cervix treated with celecoxib vs placebo.
* Compare the toxicity of these drugs in these patients.
* Determine, preliminarily, the effect of celecoxib on cyclooxygenase-2 expression and human papilloma virus expression in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to high-grade squamous intraepithelial lesion status (cervical intraepithelial neoplasia [CIN] 2 vs CIN 3). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral celecoxib twice daily for 1 month.
* Arm II: Patients receive oral placebo twice daily for 1 month. In both arms, treatment repeats monthly for 3 courses in the absence of disease progression or unacceptable toxicity. All patients then undergo loop electrosurgical excision procedure or cone biopsy to determine response.

PROJECTED ACCRUAL: A total of 100 patients (50 per treatment arm) will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed high-grade squamous intraepithelial lesions (HGSIL) of the cervix
* Cervical intraepithelial neoplasia (CIN) 2 (moderate dysplasia) OR CIN 3 (severe dysplasia, carcinoma in situ)
* Must have remaining HGSIL after biopsy
* No suspicion of invasive cancer by colposcopy within the past 28 days
* No invasive or preinvasive high-grade intraepithelial neoplasia by endocervical curettage within the past 56 days

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* SGOT and SGPT less than 2.0 times upper limit of normal (ULN)
* Bilirubin less than 2.0 times ULN

Renal

* Creatinine less than 2.0 mg/dL

Immunologic

* No prior asthma, urticaria, or allergic-type reactions to aspirin or other NSAIDs
* No allergy to sulfonamides
* No known sensitivity to celecoxib
* No known AIDS or HIV-associated complex

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or adequately treated stage I or II cancer currently in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* No prior pelvic radiotherapy

Surgery

* See Disease Characteristics

Other

* More than 3 months since prior topical medications for genital condyloma
* No prior treatment for squamous intraepithelial lesions
* No concurrent topical medications for genital condyloma
* No other concurrent treatment
* No concurrent chronic (daily for more than 30 days) aspirin
* No other concurrent nonsteroidal anti-inflammatory drugs (NSAIDs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William R. Robinson, MD, Study Chair — Harrington Cancer Center